CLINICAL TRIAL: NCT03583905
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-330 and D086 Combination Therapy in Hypertensive Patients With Dyslipidemia
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-333 Tablet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 170HT/DL17007
Record Dates: First submitted 2018-05-24; First posted 2018-07-12 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-04

CONDITIONS: Hypertensive Patients With Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): Patients assigned to this group are treated with CKD-330, D086
  Interventions: Drug: CKD-330; Drug: D086; Drug: Placebo of D723
- Placebo Group 1 (Placebo Comparator): Patients assigned to this group are treated with 1 Placebo Tab.(Placebo of the D086)
  Interventions: Drug: CKD-330; Drug: Placebo of D086; Drug: Placebo of D723
- Placebo Group 2 (Placebo Comparator): Patients assigned to this group are treated with 1 Placebo Tab.(Placebo of the CKD-330)
  Interventions: Drug: Placebo of CKD-330; Drug: D086; Drug: D723

INTERVENTIONS:
Drug: CKD-330 — CKD-330 Tab.
  Arms: Experimental Group 1; Placebo Group 1
Drug: Placebo of CKD-330 — Placebo of CKD-330 Tab.
  Arms: Placebo Group 2
Drug: D086 — D086 Tab.
  Arms: Experimental Group 1; Placebo Group 2
Drug: Placebo of D086 — Placebo of D086 Tab.
  Arms: Placebo Group 1
Drug: D723 — D723 Tab.
  Arms: Placebo Group 2
Drug: Placebo of D723 — Placebo of D723 Tab.
  Arms: Experimental Group 1; Placebo Group 1

SUMMARY:
To Evaluate the Efficacy and Safety of CKD-333

DETAILED DESCRIPTION:
A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-330 and D086 Combination Therapy in Hypertensive Patients with Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a mean sitting systolic blood pressure (MSSBP) ≥ 140 mmHg measured on selected arms after run-in period
2. Lipid levels measured after run-in period were:

   * Group 1: hypertension + dyslipidemia only → fasting LDL-C ≥ 160 mg / dL
   * Group 2: hypertension + dyslipidemia + cardiovascular risk factor more than 1 → fasting LDL-C ≥ 130mg / dL
   * Group 3: hypertension + dyslipidemia + coronary artery disease or equivalent or 10-year risk assessed by Framingham Point Score greater than 20% → fasting LDL-C ≥ 100 mg / dL

Exclusion Criteria:

1. Patients whose blood pressures measured at Visit 2 were:

   * Patients with MSSBP ≥ 180 mmHg and / or MSDBP ≥ 110 mmHg
2. Patients who had lipid levels measured at Visit 2

   * Patients with fasting LDL-C <100 mg / dL or fasting LDL-C> 250 mg / dL and / or TG ≥ 500 mg / dL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change rate from baseline in LDL-C | 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Change from baseline in MSSBP | 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 2

SECONDARY OUTCOMES:
Change rate from baseline in LDL-C | 4 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Change from baseline in LDL-C | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Attainment of LDL-C treatment goal as defined by NCEP ATP Ⅲ Guideline | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Change from baseline in MSSBP(mmHg) | 4 weeks after drug administrations
  Compare experimental group 1 with placebo group 2
Change from baseline in MSDBP | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 2
Attainment of normal blood pressure as defined by JNC Ⅶ | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 2
Change from baseline in TC | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Change from baseline in TG | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
Change from baseline in HDL-C | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
change rate from baseline in TC | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
change rate from baseline in TG | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1
change rate from baseline in HDL-C | 4, 8 weeks after drug administrations
  Compare experimental group 1 with placebo group 1

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Catholic University Seoul St. Mary's Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Yonsei University Medical Center Gangnam Severance Hospital, Seoul
  - Yonsei University Medical Center Severance Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No